CLINICAL TRIAL: NCT07094061
Title: Neurobehavioral Signatures of Sign- and Goal-Tracking in Emerging Adults: Translation of a Preclinical Model
Acronym: SIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lora Cope, Assistant Professor Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00269332; R01DA058010 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Substance Use; Healthy
Keywords: Functional magnetic resonance imaging (fMRI); Questionnaires; Interviews; Behavioral tasks
MeSH Terms: conditions — Substance-Related Disorders | interventions — Magnetic Resonance Imaging; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a longitudinal, repeated-measures, naturalistic study that will take place at the University of Michigan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment group (Experimental)
  Interventions: Device: fMRI; Behavioral: Questionnaires and surveys; Behavioral: Behavioral tasks and eye tracking

INTERVENTIONS:
Device: fMRI — Participants will have an MRI to scan participants brains and will wear skin conductance electrodes on the hand and fill out questionnaires. Scanning will take approximately 90 minutes. While lying in the scanner, participants will be asked to perform some tasks. The tasks will be presented to participants visually on a screen in the scanner and eye movements will also be tracked during some of these tasks. Participants will respond to stimuli with button presses that are recorded by computer.
Behavioral: Questionnaires and surveys — Participants will have multiple visits during this study and fill out various surveys at these visits.
Behavioral: Behavioral tasks and eye tracking — Participants will perform behavioral tasks while having eye-tracking hardware monitor participants eye movements. A video camera will be used to record eye movements during the behavioral tasks.

SUMMARY:
This study seeks to understand individual differences in personality, brain function, and behavior.

Study hypothesis:

- A stronger sign-tracking bias will be associated with a bottom-up processing style characterized by less adaptive attentional- and impulse-control as well as hyperactive reward processing, whereas a stronger goal-tracking bias will be associated with a top-down processing style characterized by strong attentional- and impulse-control as well as normative reward processing.

ELIGIBILITY:
Inclusion Criteria:

* 18-20 years old at baseline
* Right-handed
* Medically/physically able to give informed consent
* English-speaking
* Substance use is free to vary, but for participants with a history of substance use, ≥ 1 use of cannabis (including less than a full dose)

Exclusion Criteria:

* Acute or chronic medical or neurological illness (e.g., diabetes, epilepsy, migraine)
* History of psychosis in self or first-degree relative
* Current treatment for substance use disorder
* Current or past 6-month treatment with centrally acting medications (not including attention deficit hyperactivity disorder (ADHD) medication)
* Intelligence quotient (IQ) < 70
* Lifetime history of head trauma with loss of consciousness > 5 minutes
* Reliance on glasses to be able to read small text at a distance of approximately 30 inches
* Colorblindness
* MRI contraindication (e.g., pregnancy, metal implants, claustrophobia) per protocol

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between Pavlovian conditioned approach (PavCA) bias score (out-of-scanner) and composite cannabis use score | Baseline
  PavCA bias score based on eye gaze during the Pavlovian conditioned approach task will be correlated with a cannabis use composite score based on the Substance Use History and Timeline Follow-Back.

SECONDARY OUTCOMES:
Correlation between PavCA bias score (out-of-scanner) and activation from the Cannabis Cue Reactivity Task (P-CAN) | Baseline
  PavCA bias score based on eye gaze during the Pavlovian conditioned approach task will be correlated with the first principal component of average parameter estimates from the following regions extracted for the cannabis vs. neutral contrast: ventral striatum, anterior cingulate, posterior cingulate, insula, amygdala, orbitofrontal cortex, inferior occipital cortex, and inferior parietal cortex

CONTACTS AND LOCATIONS:
Overall Officials: Lora Cope, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Rachel Upjohn Building, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The scientific data collected will be preserved to enable sharing via Inter-university Consortium for Political and Social Research (ICPSR)/National Addiction & HIV Data Archive Program (NAHDAP). The demographic, clinical, and psychometric raw and composite data will both be preserved and shared, and respondent identifiers will be removed and maintained in a secure file for future contact purposes.
  Where applicable, sensitive data will be managed using ICPSR/NAHDAP's restricted data dissemination practices to ensure the data are kept confidential.
Supporting Information: Study Protocol, ICF
Time Frame: The investigator/project team will contact ICPSR/NAHDAP 3-4 months before the required release date to determine if there would be lag time between data submission and ICPSR/NAHDAP's release of the data. ICPSR/NAHDAP permanently archives deposited files, supporting the data through changing technologies, new media, and data formats.
Access Criteria: The only requirements to access downloadable, de-identified data through ICPSR/NAHDAP are user registration and agreement to ICPSR/NAHDAP's Terms of Use, which require users to agree to not re-disseminate data, to use appropriate data citation, and to maintain human subjects protections. In the case of restricted-use, sensitive data, ICPSR/NAHDAP requires an application to access the data. As part of the application process, the data user's institution must enter into a Restricted Data Use Agreement with ICPSR/NAHDAP among other application components and data security requirements. Restricted data users are approved to access the data for a limited time period and in a controlled environment through the Virtual Data Enclave or a local computing environment that they secure themselves.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/index.html